CLINICAL TRIAL: NCT03348540
Title: Randomized Clinical Trial of Attention Control Training for Symptoms of PTSD in Children
Brief Title: Attention Control Training for PTSD in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Amy Badura Brack, Professor of Psychology, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1123267
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control Training (Experimental): * 6 sessions in the clinic lasting approximately 10 minutes each.
  * Each session will consist of 128 presentations of pairs of neutral and threatening stimuli, followed by the presentation of a response cue (right or left arrow to be clicked on a computer keyboard).
  Interventions: Behavioral: Attention Control Training
- Comparison Task (Placebo Comparator): 6 sessions in the clinic of a presumably inactive neutral-neutral stimuli intervention lasting approximately 10 minutes each.
  • Each session will consist of 128 presentations of pairs of faces, followed by the presentation of a response cue (right or left arrow to be clicked on a computer keyboard).
  Interventions: Behavioral: Comparison Task

INTERVENTIONS:
Behavioral: Attention Control Training — Attention control training teaches participants that the emotional salience of cues (i.e., threatening or neutral) is not related to successful completion of the computerized response task, and thus, teaches participants to ignore irrelevant threat-related contingencies (Badura-Brack et al., 2015).
  Arms: Attention Control Training
Behavioral: Comparison Task — Neutral- neutral stimuli prior to response task
  Arms: Comparison Task

SUMMARY:
Participants will complete a pre and post training psychological assessment. Participants will be assigned to attention control training or the comparison stimuli computer task in a double-blind randomized control trial design. Both computerized dot probe tasks display two faces on a computer screen, one above the other, followed by a small right or left arrow appearing in the location vacated by one of the faces. Participants are required to respond as quickly as they can by pressing the indicated right or left arrow on their computer keyboard without compromising accuracy. Participants complete 6 training sessions.

ELIGIBILITY:
Inclusion Criteria:

* significant symptoms of PTSD and qualifying traumatic event

Exclusion Criteria:

* new traumatic event within one month of beginning the trial

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Change in posttraumatic stress disorder (PTSD) symptoms from pre to post test | 10 minute long administration, given twice to measure change scores from pre and post training approximately 1 month apart
  PTSD self-report questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton Univeristy, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Badura-Brack AS, Naim R, Ryan TJ, Levy O, Abend R, Khanna MM, McDermott TJ, Pine DS, Bar-Haim Y. Effect of Attention Training on Attention Bias Variability and PTSD Symptoms: Randomized Controlled Trials in Israeli and U.S. Combat Veterans. Am J Psychiatry. 2015 Dec;172(12):1233-41. doi: 10.1176/appi.ajp.2015.14121578. Epub 2015 Jul 24. PMID 26206075